#### The GlaxoSmithKline group of companies

| Division | · | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for Study 201840: An Exploratory Randomized, 2-Part, Single-blind, 2-Period Crossover Study Comparing the Effect of Albiglutide with Exenatide on Regional Brain Activity Related to Nausea in Healthy Volunteers

Compound Number : GSK716155

Effective Date : [20-Nov-2017]

### **Description:**

- The purpose of this RAP is to describe the planned analyses and outputs that will be reported by GSK Clinical Statistics & Programming Department.
- This RAP is to describe Part A only since the study was terminated early and Part B was cancelled prior to the completion of Part A; however, Part A was completed as planned.
- Analyses that will be performed by Massachusetts General Hospital (MGH)/Health Science & Technology (HST) Athinoula A. Martinos Center for Biomedical Imaging [Martinos] are described separately and are provide in Attachment 11.

#### **Author's Name and Functional Area:**

| PPD | 20-Nov-2017 |
|----------------------------------------------|--------------|
| Principle Statistician (Clinical Statistics) | 20-1107-2017 |

### Approved by:

| PPD | 30-Nov-2017 |
|--------------------------------|--------------|
| Director (Clinical Statistics) | 30-1NOV-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMM<br>2.1. | | KEY PROTOCOL INFORMATIONs to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | ojective(s) and Endpoint(s) | |
| | 2.3. | | esign | |
| | 2.4. | | al Hypotheses | |
| 3. | | | LYSES | |
| | 3.1.<br>3.2. | | alysesalyses | |
| 4. | | | PULATIONS | |
| | 4.1. | | Deviations | 9 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | 10 |
| 6. | | | ATION ANALYSES | |
| 0. | 6.1. | | v of Planned Analyses | |
| | 6.2. | Demogra | aphic and Baseline Characteristics | 11 |
| | 6.3. | Exposure | e to Study Drug | 11 |
| | 6.4. | Medicati | ons | 12 |
| 7. | PRIMA<br>7.1. | | FISTICAL ANALYSESAnalyses | |
| | 7.1. | 7.1.1. | | |
| | | | · | |
| 8. | | | STATISTICAL ANALYSES | |
| | 8.1. | | ry Efficacy Analyses | |
| | 8.2. | 8.2.1. | Tolerability Analyses Overview of Planned Analyses | |
| | | 8.2.2. | Vital Signs | |
| | | 8.2.3. | Clinical Laboratory Evaluations | |
| | | 8.2.4. | Adverse Events | |
| | | 8.2.5. | Most Common Adverse Events | - |
| | | 8.2.6. | Deaths and Serious Adverse Events | |
| | | 8.2.7. | Nausea Rating Scale | |
| | | 8.2.8. | GI VAS | |
| | | 8.2.9. | MSAQ | |
| | | 8.2.10. | Pregnancies | |
| 9. | REFE | RENCES. | | 17 |
| 10. | | | . 4. Destacel Desisting Management and Definitions for | 18 |
| | 10.1. | | x 1: Protocol Deviation Management and Definitions for | 10 |
| | 10.2. | | ocol Populationx 2: Time & Events | |
| | 10.2. | | Protocol Defined Time & Events | |

### **CONFIDENTIAL**

| | 10.3. | Appendix 3: Assessment Windows | 21 |
|-----|-------|-------------------------------------------------------|----|
| | | 10.3.1. Definitions of Study Day | 21 |
| | 10.4. | | 22 |
| | | 10.4.1. Laboratory | |
| | | 10.4.2. Vital Signs | |
| | 10.5. | <b>G</b> | |
| | | 10.5.1. Study Treatment Display Descriptors | |
| | 10.6. | Appendix 6 – Abbreviations & Trade Marks | 26 |
| | | 10.6.1. Abbreviations | |
| | | 10.6.2. Trademarks | 27 |
| | 10.7. | | |
| | | 10.7.1. Data Display Numbering | 28 |
| | | 10.7.2. Study Population Tables | 29 |
| | | 10.7.3. Efficacy Tables | |
| | | 10.7.4. Safety Tables | |
| | | 10.7.5. ICH Listings | 30 |
| | | 10.7.6. Non-ICH Listings | 31 |
| 11. | ATTA | CHMENTS [DOCUMENTATION FROM MARTINOS] | 32 |
| | | Reporting & Analysis Plan for Imaging Data for Part A | |
| | | 11.1.1 Overview of Quality Control for Imaging Data | 32 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this RAP is to describe the planned analyses and outputs that will be reported by GSK Clinical Statistics & Programming Department. At the time of the RAP preparation, the study had terminated early and Part B was cancelled prior to the completion of Part A; however, Part A was completed as planned. This RAP is for Part A only. |
| | Analysis that will be performed by Massachusetts General Hospital (MGH)/Health Science & Technology (HST) Athinoula A. Martinos Center for Biomedical Imaging [Martinos] is described in a separate document added as Attachment 11 to this RAP. |
| Protocol | This RAP is based on protocol amendment 1 [(Dated: 28/Nov/2016) of study GSK 201840 (GSK Document No.: 2015N250344_02] and eCRF Version 5.1. |
| Primary<br>Objective | <ul> <li>To explore the effect of single dose 50 mg albiglutide compared to single dose<br/>10 µg exenatide on regional brain activity and connectivity associated with<br/>nausea in healthy volunteers</li> </ul> |
| Primary | Resting-state BOLD signal (fMRI) |
| Endpoints | Regional cerebral blood flow (rCBF) (fMRI-ASL) |
| | Glutamate concentration in nausea-associated brain regions (MRS) |
| | GABA concentration in nausea-associated brain regions (MRS) |
| Study<br>Design | This is a phase IV, 2-part, 2-period crossover, single dose, randomized, single blind (blinded to both the subject and the imaging evaluators analysing the MRI data), placebo and active-controlled study in adult healthy volunteers who are susceptible to motion sickness. |
| Planned<br>Analyses | <ul> <li>Analysis of primary and some secondary endpoints for Part A will be performed<br/>by Martinos. Details are described in <u>Attachment 11</u>.</li> </ul> |
| Analysis<br>Populations | For this study, the analysis set will include subjects who have valid data as determined at the discretion by the imaging laboratory. |
| Hypothesis | No primary hypothesis was pre-specified due to the exploratory nature of the study. |
| Primary<br>Analyses | The primary analyses will be exploratory in nature and will consist of summary outputs and listings and will cover the following primary endpoints: |
| Resting-state BOLD signal (fMRI) | |
| | Regional cerebral blood flow (rCBF) (fMRI-ASL) |
| | Glutamate concentration in nausea-associated brain regions (Magnetic resonance spectroscopy (MRS)) |

| Overview | Key Elements of the RAP |
|---|---|
| | GABA concentration in nausea-associated brain regions (MRS) |
| Secondary<br>Analyses | Secondary analyses will also be exploratory in nature and will consist of summary statistics and listings for the following endpoints: |
| | 1. Heart rate** |
| | 2. heart rate variability** |
| | 3. respiratory rate** |
| | 4. ECG intervals** |
| | 5. blood pressure** |
| | 6. skin conductance level** |
| | Secondary analyses consisting of summary statistics for continuous variables and frequency and percent for categorical variables will be performed for the following safety endpoints: |
| | 1. Vital signs |
| | 2. clinical laboratory tests* |
| | 3. adverse events |
| | 4. Nausea ratings scale ** |
| | 5. Gastrointestinal-Visual analogue scale (Gl VAS) |
| | 6. Motion Sickness Assessment Questionnaire (MSAQ) |
| | *Only listings will be provided. |
| | ** Will be provided by Martinos |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Since the study was terminated early; Part B was cancelled prior to the completion of Part A, 4 subjects completed Part A as planned and a decision was made to not complete group analysis of the 4 subjects. Therefore, no interim analyses will be performed as stated in the originally planned statistical analysis specified in the protocol / protocol amendment 1 [(Dated: 28/Nov/2016)].

# 2.2. Study Objective(s) and Endpoint(s)

| Ok | pjectives | En | dpoints |
|---|---|---|---|
| Pr | Primary Objectives | | mary Endpoints |
| To explore the effect of single dose 50 mg albiglutide compared to single dose 10 g exenatide on regional brain activity and connectivity associated with nausea in healthy volunteers | | <ul> <li>Resting-state BOLD signal (fMRI)</li> <li>Regional cerebral blood flow (rCBF) (fMRI-ASL)</li> <li>Glutamate concentration in nausea-associated brain regions (MRS)</li> <li>GABA concentration in nausea-associated brain regions (MRS)</li> </ul> | |
| Se | condary Objectives | Se | condary Endpoints |
| • | To evaluate autonomic effects of single dose 50 mg albiglutide compared to single dose 10 lg exenatide | • | Heart rate, heart rate variability, respiratory rate, ECG intervals, blood pressure, skin conductance level |
| • | To assess safety and tolerability of single dose 50 mg albiglutide and single dose 10 lg exenatide | • | Vital signs, clinical laboratory tests, adverse events,<br>Nausea ratings scale, GI VAS, and MSAQ |
| Ex | ploratory Objectives | Ex | ploratory Endpoints |
| • | To evaluate gastric myoelectrical activity (GMA) of single dose 50 mg albiglutide compared to single dose10 lg exenatide | • | GMA: Dominant power (DP), Dominant frequency (DF), % time spent in 3 frequency bands (Bradygastria, Normal, Tachygastria) and Ratio of power in post-task versus pretask. (Martinos will provide analysis data if considered valid) |

### 2.3. Study Design



# 2.4. Statistical Hypotheses

No primary hypothesis was pre-specified due to the exploratory nature of the study.

### 3. PLANNED ANALYSES

### 3.1. Interim Analyses

No interim analyses will be performed since the study was terminated early and Part B cancelled prior to the completion of Part A; however, Part A was completed as planned.

## 3.2. Final Analyses

The final reporting will be performed after the completion of the following sequential steps:

- 1. All subjects have completed Part A of the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared.

The reporting and analysis of imaging data after completion of the study will be performed by Martinos. Details are described in <a href="Attachment 11"><u>Attachment 11</u></a>.

### 4. ANALYSIS POPULATIONS

| Population Definition / Criteria | | Analyses Evaluated |
|---|---|---|
| All Screened | All participants who were screened will be considered for this population. This population will be used for summarizing screening status | Screen failure |
| Enrolled | All participants who were successfully screened<br>and enrolled for the trial and for whom a record<br>exists on the study database. | Study population |
| Safety | <ul> <li>Comprise of all subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> <li>This population will include subjects who were replaced due to imaging data being invalid or not evaluable but received study drug.</li> </ul> | Safety |
| Analysis Set (Randomised) | <ul> <li>Comprise of all randomized subjects who receive treatment and with valid imaging data, that will be determined by Martinos.</li> <li>Subjects who are replaced are excluded from this population.</li> </ul> | Imaging (Mechanism of Action) |

#### NOTES:

• Please refer to Appendix 7: List of Data Displays which details the population to be used for each display being generated.

### 4.1. Protocol Deviations

• Protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be reviewed and tracked throughout the conduct of the study. However, there is no perprotocol analysis that will be performed for this study.

Only listings of the Protocol deviations will be provided if any.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Imaging Analysis Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Values of Potential Clinical Importance |
| Error!<br>Referen | : Data Display Standards & Handling Conventions |
| ce<br>source<br>not<br>found. | |
| Error!<br>Referen | : Abbreviations & Trade Marks |
| ce<br>source<br>not<br>found. | |
| Error!<br>Referen<br>ce<br>source<br>not<br>found. | : List of Data Displays |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population summary will be based on the Safety population, unless otherwise specified.

Subject characteristics and safety data (captured in the eCRF) will be reported by GSK. GSK Statistics & Programming (S&P) will provide summary tables data listings of subject characteristics and safety data for Part A.

Table 2 provides an overview of the planned study population summaries, with full details of data displays being presented in Appendix 7: List of Data Displays.

Table 2 Overview of Planned Study Population Summaries

| [Endpoint / Parameter / Display Type] | Data | Data Displays Generated | |
|---|---|---|---|
| | Table | Figure | Listing |
| Part A | | | |
| Reasons for Screening Failures | Υ | | Υ |
| Randomization | | | Υ |
| Subject Disposition | Υ | | Υ |
| Summary of Number of Subjects by Site ID | Y | | |
| Demographics and Baseline Characteristics | Y | | Y |
| Race (& Racial Combinations) | Y | | Y |
| Age Ranges | Y | | |
| Medical Condition & Concomitant Medications | | | |
| Medical History | | | Y |
| Concomitant Medication | | | Y |
| Exposure | | | |
| Exposure to Study Drug | | | Y |

#### NOTES:

# 6.2. Demographic and Baseline Characteristics

Continuous variables such as age, body mass index, weight, and height will be summarized using descriptive statistics (n, mean, standard deviation, and median, minimum, maximum). Categorical variables including sex, race, ethnicity, tobacco use, alcohol intake, caffeine intake, and baseline weight category (<90 kg or ≥90 kg) will be summarized using numbers and percentages.

Continuous variables such as age, body mass index, weight, and height will be presented in a by-subject listing. Listings will be presented using the safety population.

# 6.3. Exposure to Study Drug

<sup>•</sup> Y = Yes display generated.

A by-subject listing of study drug administration will also be presented.

## 6.4. Medications

Any prior and concomitant medication used during the study will be recorded and coded using GSKDrug Dictionary (GSKDRUG), which will be updated whenever available throughout the life of the study.

Any medication used during the study will be recorded, which will be updated whenever available throughout the life of the study.

All medications will be listed.

## 7. PRIMARY STATISTICAL ANALYSES

The imaging data will be reported by Martinos at the end of the study. Details of the planned analyses are described in <u>Attachment 11</u>.

# 7.1. Efficacy Analyses

### 7.1.1. Overview of Planned Efficacy Analyses

The primary efficacy analyses will be based on the all randomised population, unless otherwise specified.

The efficacy analyses will be performed by Martinos, details of the planned analysed are described in Attachment 11.

# 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Secondary Efficacy Analyses

The secondary analysis to list autonomic effects of albiglutide compared to exenatide will be performed and reported by Martinos. Details of the planned analyses are described in <a href="https://doi.org/10.2016/j.jep-10.2016/

### 8.2. Safety & Tolerability Analyses

### 8.2.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Safety data (captured in the eCRF) will be reported by GSK. GSK Statistics & Programming (S&P) will provide summary tables and data listings of safety data for Part A data.

Table provides an overview of the planned analyses, with further details of data displays being presented in Appendix 7: List of Data Displays.

Table 3 Overview of Planned Safety & Tolerability Analyses

| [Endpoint / Parameter/ Display | Data Displays Generated | | | |
|---|---|---|---|---|
| Type] | Summary | | Individual | |
| | Table | Figure | Figure | Listing |
| Vital Signs | Υ | | | Υ |
| Clinical Laboratory* | | | | Υ |
| Adverse Events | Υ | | | Υ |
| 12-lead ECG | | | | Υ |
| GI- VAS | Υ | | | Υ |
| MSAQ | Υ | | | Υ |
| MRI | | | | Y |

<sup>\*</sup>Clinical Laboratory will include Fasting Plasma Glucose.

### 8.2.2. Vital Signs

The vital sign summary and analysis will include systolic blood pressure (mmHg), diastolic blood pressure (mmHg), and heart rate (bpm).

For Part A, each vital sign parameter at every scheduled assessment time point will be summarized using descriptive statistics. Additionally, the number of subjects with vital signs of potential clinical concern will also be summarized. The criteria for vital signs of potential clinical concern are detailed in Appendix 7: Values of Potential Clinical Importance.

All summaries will be done for the safety population and all vital sign data will be listed.

## 8.2.3. Clinical Laboratory Evaluations

Laboratory parameters include the following tests: hematology, chemistry and urinalysis. Established or generally acknowledged methods, normal ranges, and quality control procedures will be supplied by Quest Diagnostics Clinical Laboratory for the study records.

All laboratory parameters as collected will be presented in by-subject listings at every scheduled assessment time point for the safety population.

Additionally, listing of the number of subjects with laboratory values of potential clinical concern will be provided and scheduled assessment time point for hematology and chemistry. The criteria for laboratory values of potential clinical concern are detailed in Appendix 7: Values of Potential Clinical Importance.

Listings of clinical laboratory evaluations will be provided.

#### 8.2.4. Adverse Events

All AEs will be coded using MedDRA which will be updated whenever available throughout the life of the study.

For Part A safety review, adverse events will be summarized by treatment group. Summary of the number and percentage of subjects with any AE and the total number of AEs recorded will be provided. SAEs will be summarized.

All AEs will be listed in a subject data listing.

#### 8.2.5. Most Common Adverse Events

A summary of most common adverse events (>2% total incidence in any treatment arm) by treatment will be produced.

#### 8.2.6. Deaths and Serious Adverse Events

Deaths and serious adverse events will be listed.

### 8.2.7. Nausea Rating Scale

Nausea rating scale will be provided by Martinos.

#### 8.2.8. GI VAS

Summary statistics outputs and listings for GI VAS will be provided

#### 8.2.9. MSAQ

Summary statistics outputs and listing for MSAQ will be provided.

#### 8.2.10. Pregnancies

Listings for Pregnancies will be produced if any.

# 9. REFERENCES

None.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Values of Potential Clinical Importance |
| Section | <ul> <li>: Data Display Standards &amp; Handling Conventions</li> <li>Study Treatment &amp; Sub-group Display Descriptors</li> </ul> |
| Section 10.6 | Appendix 6: Abbreviations & Trade Marks |
| Section 10.7 | Appendix 7: List of Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per-Protocol Population

The Protocol Deviation Management Plan (21/Feb/2017) will be used to identify the important protocol deviations. It is intended to categorize important protocol deviations that are anticipated to occur in a study and to document study-specific requirements for cross-functional team review of these protocol deviations and other deviations that may occur in the study. There is no pre-defined per protocol population criteria.

#### 10.2. **Appendix 2: Time & Events**

#### 10.2.1. **Protocol Defined Time & Events**

| | Scree | | | | | | S | essi | on 1 | | | | | | Wash<br>out | | | | Ses | sion | 2 | | | F/<br>U |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5 | | | Da | y 1 | | | | | Da | ıy 8± | :1 <sup>m</sup> | | | | | | | D | ay 4: | ±1 <sup>m</sup> | | | |
| Procedure | Week -4 to -1 | | Pre-MRI | MRI | М | ost<br>RI | Day 5±1™ | -2 h | -0.5 h | 0 h | 0.5 h | 1 h | M | ost<br>IRI | 6-9 weeks | Day 1 | -2 h | -0.5 h | 0 h | 0.5 h | 1 h | P<br>M | ost<br>IRI | Week |
| | p -7 | | MR! | 고 | 0.5 h | 1 | m<br>H | Ъ | 5 h | ъ | 5 h | 5 | 0.5 h | 1 h | eeks | _ | Ъ | 5 h | 5 | 5 h | ъ | 0.5 h | 1 h | 13 |
| Visit (all out-patient) | 1 | 2 | | . ; | 3 | | 4 | | | | 5 | | | | | 6 | | | | 7 | | | | 8 |
| Informed Consent | X | | | | | | | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | | | | | | | |
| Medical history <sup>a</sup> | X | | | | | | | | | | | | | | | | | | | | | | | |
| Prior/Concomitant medication <sup>b</sup> | Х | Х | Х | | | | Х | Х | | | | | | | | Х | Х | | | | | | | Х |
| Complete physical | Х | | | | | | | | | | | | | | | | | | | | | | | |
| Brief physical | | | | | | | | Х | | | | | | | | | Х | | | | | | | Х |
| Vital signs | X | Х | Χ | | Χ | | Х | Х | | | | | Х | Χ | | Χ | Χ | | | | | Χ | Х | X |
| Urine Drug, Breath Alcohol/Cotinine | X | X | Χ | | | | Х | X | | | | | | | | Χ | Χ | | | | | | | |
| 12-lead ECG <sup>e</sup> | X | | | | | | | | | | | | | | | | | | | | | | | |
| Pregnancy test (WCBP) <sup>c</sup> | X | | Х | | | | | | | | | | | | | Χ | | | | | | | | Х |
| HIV, Hep B and Hep C screen <sup>d</sup> | X | | | | | | | | | | | | | | | | | | | | | | | |
| Clinical laboratory tests <sup>e</sup> | Х | | | | | | | | | | | | | | | Χ | | | | | | | | |
| TSH, free T4, triglycerides, amylase | Х | | | | | | | | | | | | | | | | | | | | | | | |
| and lipase | | | | | | | | | | | | | | | | | | | | | | | | |
| Edinburgh Handedness Inventory | X | | | | | | | | | | | | | | | | | | | | | | | |
| MSSQ-short | X | | | | | | | | | | | | | | | | | | | | | | | |
| Mock fMRI <sup>±</sup> | | Х | | | | | | | | | | | | | | | | | | | | | | |

| | Scree ing | | | | | | S | essio | on 1 | | | | | | Wash<br>out | | | | Ses | sion | 2 | | | F/<br>U | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 5 | | | Da | y 1 | | | | | Da | y 8± | 1 <sup>m</sup> | | | | | Day 4±1 <sup>m</sup> | | | | | | | | | |
| Procedure | Week - | veek - | keek - | Week -4 to -1 | éek - | Pre | N | Po<br>M | ost<br>RI | Day 5 | 45 | -0.5 | 0 | 0. | _ | | ost<br>IRI | 6-9 v | Day | d's | -0.5 | 0 | 0.5 | 1 | ost<br>IRI | Week |
| | to -1 | | Pre-MRI | MRI | 0.5 h | 1<br>h | 5±1m | -2 h | 5 h | 0 h<br>0.5 h | 0.5 h | 1<br>h | 0.5 h | 1<br>h | 6-9 weeks | 1 | -2 h | 5 h | 0 h | 5 h | ь | 0.5 h | <u></u> | 13 | | |
| Randomization | | Х | | | | | | | | | | | | | | | | | | | | | | | | |
| Dosing albiglutide or placebo <sup>g</sup> | | | | | | | Х | | | | | | | | | Х | | | | | | | | | | |
| Dosing exenatide or placebo <sup>g</sup> | | | | | | | | | | Χ | | | | | | | | | Х | | | | | | | |
| MRI <sup>h</sup> | | | | Χ | | | | | | | | Χ | | | | | | | | | Х | | | | | |
| Autonomic monitoring | | | | Χ | | | | | | | | Χ | | | | | | | | | Х | | | | | |
| Electrogastrogram | | | | Χ | | | | | | | | Χ | | | | | | | | | Х | | | | | |
| VAS | | | Х | | Х | | | | | | Х | | Х | | | | | | | Х | | Х | | | | |
| MSAQ <sup>i</sup> | | | | | Х | | | | | | | | Х | | | | | | | | | Х | | | | |
| Capillary blood glucose | | | | | | | | | | | | | Х | | | | | | | | | Х | | | | |
| Fasting Plasma Glucose | | | | | | | | | | | | | Χ | | | | | | | | | Х | | | | |
| Snack <sup>j</sup> | | | | | Χ | | | | | | | | Χ | | | | | | | | | Х | | | | |
| AE assessment <sup>k</sup> | | | <== | | | ==> | < | | | | | | | > | | < | | | | | | | -> | X | | |
| Discharge <sup>1</sup> | | | | | | Χ | | | | | | | | Х | | | | | | | | | X | | | |

- a. Medical history includes alcohol/tobacco/caffeine usage.
   b. Prior-Medications are defined as prescription or over-the counter medications taken within 30 days of Screening. Record concomitant medications and or changes.
   c. WCBP is women of child-bearing potential. Serum pregnancy test at Screening. Urine pregnancy at other specified time points.
   d. If test otherwise performed within 1 month prior to first dose of study treatment, testing at screening is not required.
   e. See Table 2 for list of laboratory parameters. Unscheduled Safety Labs and ECGs can be done at any time if the Investigator considers the assessments appropriate for subject safety.

  f. Mock fMRI is performed on a separate day during the screening period. Scheduling should allow at least 1 week between the Mock fMRI and the next MRI scan.

- g. Albiglutide, exenatide or placebo is administered according to randomization sequence.
  h. All MRI include resting-state fMRI, ASL and MRS. Off-therapy MRI scan includes visual nauseogenic task fMRI and can be initiated once -assessments are completed. The on-therapy scan should be initiated 1 hr ±15min post the exenatide or exenatide placebo dose. Pre-scan procedure timings are suggested times to allow completion of activities. Post MRI procedure should be completed at the noted times ±15 min.

Note: reference to Table 2 in footnote e is in the protocol.

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Definitions of Study Day

When study day is used for display or in comparisons the following algorithm will be used:

- Study day = date of assessment date of first dose + 1, if day of assessment >= first dose date
- Study day = date of assessment date of first dose, if day of assessment < first dose date

Note that the date of first dose is Day 1 and the day before the date of first dose is Day -1 (there is no Day 0).

# 10.4. Appendix 4: Values of Potential Clinical Importance

# 10.4.1. Laboratory

| | | Hematology | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Basophils | GI/L | None | None |
| Eosinophils | GI/L | None | None |
| Hematocrit | 1 | >0.1 decrease | >0.05 below LLN<br>>0.04 above ULN |
| Hemoglobin | g/L | >25 g/L decrease | >20 g/L below LLN<br>>10 g/L above ULN |
| Lymphocytes | GI/L | None | <0.5 x LLN |
| Monocytes | GI/L | None | None |
| Neutrophils | GI/L | None | <1 GI/L |
| Neutrophil<br>Bands | GI/L | None | None |
| Platelets | GI/L | None | <80 GI/L<br>>500 GI/L |
| Red Blood Cell<br>Count | TI/L | None | None |
| Segmented<br>Neutrophils | GI/L | None | <0.5 x LLN |
| White Blood Cell<br>Count | GI/L | None | >1 GI/L below LLN<br>>5 GI/L above ULN |

| | | Chemistry | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Albumin | g/L | None | >5 g/L above ULN or below LLN |
| Alkaline<br>Phosphatase | U/L | None | >3 x ULN |
| ALT | U/L | None | >3 x ULN |
| AST | U/L | None | >3 x ULN |
| Bicarbonate<br>(Carbon Dioxide<br>Content) | mmol/L | None | <16 mmol/L<br>> 40 mmol/L |
| Blood Urea | mmol/L | None | >2 x ULN |

| | | Chemistry | |
|---|---|---|---|
| Laboratory<br>Test | Units | Change from Baseline of<br>Potential Clinical Concern | Potential Clinical Concern<br>Value |
| Nitrogen | | | |
| Calcitonin | pmol/L | None | >100 |
| Calcium | mmol/L | None | <1.8 mmol/L |
| | | | >3.0 mmol/L |
| Chloride | mmol/L | None | None |
| Creatinine | umol/L | None | >159 umol/L |
| Direct Bilirubin | umol/L | None | >1.35 x ULN |
| Gamma<br>Glutamyl<br>Transferase | U/L | None | >3 x ULN |
| Glucose<br>(fasting) | mmol/L | None | <3 mmol/L<br>>22 mmol/L |
| Potassium | mmol/L | None | >0.5 mmol/L below LLN<br>>1.0 mmol/L above ULN |
| Sodium | mmol/L | None | >5 mmol/L above ULN or below LLN |
| Total Bilirubin | umol/L | None | >1.5 x ULN |
| Total Protein | g/L | None | >15 g/L above ULN or below LLN |
| Uric acid | umol/L | None | >654 umol/L |
| Free Fatty Acids | mmol/L | None | None |
| HDL Cholesterol | mmol/L | None | None |
| LDL Cholesterol | mmol/L | None | None |
| Triglycerides | mmol/L | None | > 9.04 mmol/L |
| Total<br>Cholesterol | mmol/L | None | None |

| Liver Function Tests | |
|----------------------|---------------------------------------------------|
| Laboratory Test | Potential Clinical Concern Value |
| ALT | ≥2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | $\geq$ 3 x ULN and Total Bilirubin $\geq$ 2 x ULN |
| AST | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |
| | $\geq$ 3 x ULN and Total Bilirubin $\geq$ 2 x ULN |
| Total Bilirubin | ≥ 1.5 x ULN |
| | ≥ 2 x ULN |
| | ≥ 3 x ULN |
| | ≥ 5 x ULN |
| | ≥8 x ULN |
| | ≥ 10 x ULN |

# 10.4.2. Vital Signs

| Parameter | Units | Potential Clinical Concern Value |
|--------------|-------|----------------------------------|
| Systolic BP | mmHg | <100 mmHg<br>>170 mmHg |
| Diastolic BP | mmHg | <50 mmHg<br>>110 mmHg |
| Heart rate | bpm | <50 bpm > 120 bpm |

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

# 10.5.1. Study Treatment Display Descriptors

The study treatment descriptors are shown below.

| | Treatment Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Repo | rting |
| Code | Description | Description | Order [1] |
| A | Albiglutide 50mg | Albiglutide 50mg | 1 |
| E | Exenatide 10mcg | Exenatide 10mcg | 2 |

# 10.6. Appendix 6 – Abbreviations & Trade Marks

# 10.6.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| BOLD | Blood oxygen Level dependent |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| fMRI | Functional magnetic resonance imaging |
| GABA | Gama-aminobutyric acid |
| GI-VAS | Gastrointestinal-Visual analogue scale |
| IA | Interim Analysis |
| ICH | International Conference on Harmonisation |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| GUI | Guidance |
| LOC | Last Observation Carries Forward |
| MMRM | Mixed Model Repeated Measures |
| MRS | Magnetic resonance spectroscopy |
| MSAQ | Motion Sickness Assessment Questionnaire |
| PCASL | Pseudo-Continuous ASL |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |

| Abbreviation | Description |
|--------------|--------------------------------------------|
| RAMOS | Randomization & Medication Ordering System |
| rCBF | Regional cerebral blood flow |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

# 10.6.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| None |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| MedDRA |

# 10.7. Appendix 7: List of Data Displays

# 10.7.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|---------------|---------|
| Study Population | 1.1 to 1.8 NA | |
| Efficacy* | | |
| Safety | 3.1 to 3.5 | NA |
| Section | Listings | |
| ICH Listings | 1 to 21 | |
| Other Listings | 22 to 24 | |

<sup>\*</sup>Will be provided by Martinos

# 10.7.2. Study Population Tables

| Study | Study Population: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Subje | ect Dispositio | 1 | | | |
| 1.1. | Safety | ES1A | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.2. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | SAC |
| Demo | ography | | | | |
| 1.3. | Safety | DM1 | Summary of Demographic Characteristics | | SAC |
| 1.4. | Enrolled | DM11 | Summary of Age Ranges | | SAC |
| 1.5. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC |
| 1.6. | Safety | DM6 | Summary of Race and Racial Combination Details | | SAC |
| 1.7. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC |
| 1.8. | Enrolled | SP1A | Summary of Study Population | | SAC |

# 10.7.3. Efficacy Tables

All Efficacy tables and listings will be provided by Martinos.

# 10.7.4. Safety Tables

| Safet | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.1. | Safety | AE16 | Summary of Serious Adverse Events by System<br>Organ Class and Preferred Term (Number of<br>Subjects and Occurrences) | | SAC |
| 3.2. | Safety | AE15 | Summary of Common (>=2%) non-serious<br>Adverse Events by System Organ Class and<br>Preferred Term (Number of Subjects and<br>Occurrences) | | SAC |
| 3.3. | Safety | | Vital Signs of Clinical Concern by Visit | | SAC |
| 3.4. | Safety | | Summary of GI- VAS | | SAC |
| 3.5. | Safety | | Summary of MSAQ | | SAC |

# 10.7.5. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1 | Safety | CP_TA1 | Listing of Randomised and Actual Treatments | | SAC |
| 2 | Safety | ES3 | Listing of Reasons for Study Withdrawal | | SAC |
| 3 | All Screened | ES7 | Listing of Reasons for Screening Failure | | SAC |
| 4 | Enrolled | SA3a | Listing of Subjects Excluded from Any Populations | | SAC |
| 5 | Safety | DV2 | Listing of Important Protocol Deviations | | SAC |
| 6 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| 7 | Safety | DM2 | Listing of Demographic Characteristics | | SAC |
| 8 | Safety | DM10 | Listing of Race | | SAC |
| 9 | Safety | EX3 | Listing of Exposure | | SAC |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 10 | Safety | AE7 | Listings of Subject Numbers for Individual Adverse Events | | SAC |
| 11 | Safety | AE9 | Listing of All Adverse Events | | SAC |
| 12 | Safety | AE9 | Listing of Serious Adverse Events | | SAC |
| 13 | Safety | AE9 | Listing of Adverse Events Leading to<br>Withdrawal from Study / Permanent<br>Discontinuation of Study Treatment | | SAC |
| 14 | Safety | AE7 | Listing of subjects who withdrew from study due to Adverse Event | | SAC |
| 15 | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data for Subjects Abnormalities of Potential Clinical Importance | | SAC |
| 16 | Safety | LB5 | Listing of Haematology Data for Subjects with Abnormalities of Potential Clinical Importance | | SAC |
| 17 | Safety | UR2b | Listing of Urinalysis Data | | SAC |
| 18 | Safety | EG3 | Listing of 12 lead ECG Values | | SAC |
| 19 | Safety | CP_VS4 | Listing of Vital Signs for Subjects with Abnormalities of Potential Clinical Importance | | SAC |
| 20 | Safety | LB5 | Listing of all Haematology Data | | SAC |
| 21 | Safety | LB5 | Listing of all Chemistry Data | | SAC |

# 10.7.6. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 22 | Analysis | | Listing of GI- VAS | | SAC |
| 23 | Analysis | | Listing of MSAQ | | SAC |
| 24 | Analysis | | Listing of MRI | | SAC |

# 11. ATTACHMENTS [DOCUMENTATION FROM MARTINOS]

### 11.1. Reporting & Analysis Plan for Imaging Data for Part A

### 11.1.1. Overview of Quality Control for Imaging Data

Quality control procedures will include visual inspection of raw brain images for presence of various artifacts, including but not limited to, aliasing, excessive distortion, Nyquist N/2 ghosting, and signal inhomogeneities. We will also assess head motion correction parameters to ensure that subjects were not moving excessively during the functional MRI (BOLD fMRI and pCASL) scans. We will evaluate 1) total translation and rotation motion, 2) relative TR-to-TR motion, 3) number of relative translations (> 0.1 mm). For pCASL data, we will calculate rCBF and ensure values within the gray matter are within normal bounds (40-60 mm/100 g tissue/min). For <sup>1</sup>H-MRS data we will assess spectra to ensure adequate SNR (Cramer–Rao lower bounds values below 40%).

We will perform single-subject level analyses and include data from (1) resting-state BOLD fMRI, (2) pseudo-continuous arterial spin labelling (pCASL), and (3) proton-density weighted magnetic resonance spectroscopy (<sup>1</sup>H-MRS).

### **Primary Outcomes/Endpoints:**

- 1. Resting-state functional connectivity (resting-state BOLD fMRI)
- 2. Regional cerebral blood flow (rCBF) (pCASL)
- 3. Glutamine/Glutamate (Glx) and GABA concentrations (<sup>1</sup>H-MRS)

### 1. Resting-state fMRI (rs-fMRI)

Resting-state BOLD signal MRI data collected at off-therapy and exenatide post-dose MRI scan sessions will be analyzed using a whole-brain seed-to-voxel approach. The seed-to-voxel driven approach will include *a priori* seed ROIs placed in brain areas subserving nausea-related processing including regions identified from our prior study (Napadow et al. Cereb Ctx 2013). These regions will include: interoceptive/sensory (insula, dACC), emotional/affective (amygdala, pgACC), and cognitive/evaluative (dlPFC/OFC) brain areas, primary visual (V1) and extrastriate cortices (area MT+/V5). Group analyses will be performed using a paired t-test (off-therapy vs. exenatide) with FSL's FLAME (FMRIB's Local Analysis of Mixed Effects).

#### 2. pCASL

pCASL data will be analysed to assess regional cerebral blood flow (rCBF) within the brain during off-therapy relative to exenatide post-dose MRI scans. Quality control of imaging data will be performed by visual inspection with adequate data denoted by mean rCBF values over the gray matter within a previously defined normal range (i.e., 40-60 mm/100 g tissue/min). In addition, all data will undergo motion and physiological noise

correction. These rCBF maps will be calculated for each subject and each scan at the single subject-level.

#### 3. <sup>1</sup>H-MRS

Magnetic resonance spectroscopy (<sup>1</sup>H-MRS) analysis will assess regional differences in glutamine/glutamate (Glx) and GABA concentrations, normalized as a ratio with creatine. MRS quantification of metabolites of interest will be based on frequency domain analysis using a Linear Combination of Model spectra (LCModel). Cramer–Rao lower bounds (CRLBs), as reported from the LCModel analysis, will be used to assess the reliability of the major metabolites and adequate SNR. CRLBs values less than 40% will be further analyzed. Metabolite maps for each subject, and each session will be calculated.

### Secondary outcomes/endpoints:

Additional analyses will be conducted for secondary outcome measures including heart rate, heart rate variability, respiratory rate, ECG intervals, blood pressure, and skin conductance level. Electrogastrogram (EGG) data will also be analysed as a secondary exploratory outcome. We will provide clean, processed physiological data in the subject/scan directories when available (secondary ANS data will not be available from every scan due to MR-induced artifacts).